CLINICAL TRIAL: NCT04265846
Title: Prospective Clinical Study of Different Intraocular Lens Implantation Designed for the Correction of Presbyopia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Sponsor
Other Study IDs: 20191129
Record Dates: First submitted 2019-11-29; First posted 2020-02-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-03

CONDITIONS: Presbyopia; Cataract Senile
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- bifocal IOL group: The cataract patients who ask for bilateral phacoemulsification and bifocal IOLs implantation.
  Interventions: Device: bifocal IOL
- mix bifocal IOL group: The cataract patients who ask for phacoemulsification and mix different bifocal IOLs implantation bilaterally
  Interventions: Device: mix bifocal IOL
- trifocal IOL group: The cataract patients who ask for bilateral phacoemulsification and trifocal IOLs implantation.
  Interventions: Device: trifocal IOL
- EDOF IOL group: The cataract patients who ask for bilateral phacoemulsification and EDOF IOLs implantation.
  Interventions: Device: EDOF IOL
- blend vision group: The cataract patients who ask for phacoemulsification and different IOLs implantation bilaterally.
  Interventions: Device: different IOLs
- monovision designed group: The cataract patients who ask for bilateral phacoemulsification and monofocal IOLs implantation with monovision designed.
  Interventions: Device: monofocal IOL
- monofocal IOL group: The cataract patients who ask for bilateral phacoemulsification and monofocal IOLs implantation with emmetropia designed.
  Interventions: Device: monofocal IOL

INTERVENTIONS:
Device: bifocal IOL — The patients will undergo bilateral phacoemulsification and bifocal IOLs implantation.
  Groups: bifocal IOL group
Device: mix bifocal IOL — The patients will undergo phacoemulsification and mix different bifocal IOLs implantation bilaterally.
  Groups: mix bifocal IOL group
Device: trifocal IOL — The patients will undergo bilateral phacoemulsification and trifocal IOLs implantation.
  Groups: trifocal IOL group
Device: EDOF IOL — The patients will undergo bilateral phacoemulsification and EDOF IOLs implantation.
  Groups: EDOF IOL group
Device: different IOLs — The patients will undergo phacoemulsification and different IOLs implantation bilaterally.
  Groups: blend vision group
Device: monofocal IOL — The patients will undergo bilateral phacoemulsification and monofocal IOLs implantation with monovision designed.
  Groups: monovision designed group
Device: monofocal IOL — The patients will undergo bilateral phacoemulsification and monofocal IOLs implantation with emmetropia designed.
  Groups: monofocal IOL group

SUMMARY:
Compare postoperative Subjective and objective visual quality and economic efficiency of different Intraocular Lens(IOLs) implantation designed for the correction of presbyopia.

DETAILED DESCRIPTION:
Compare postoperative Subjective and objective visual quality and economic efficiency of different Intraocular Lens Implantation designed for the correction of presbyopia.The subjects will undergo bilateral uneventful phacoemulsification and implantation of IOL.The subjects will be divided into several groups according to the type of the IOLs，including monofocal IOL group,monovision designed group ，bifocal IOL group, mix bifocal IOL group，trifocal IOL group，Exteded Depth of Focus(EDOF) IOL group and blend vision group. Compare the Subjective and objective visual quality and economic efficiency among these groups at 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral cataract
* Regular corneal topography and Preoperative corneal astigmatism ≤ 0.75 Diopter

Exclusion Criteria:

* Pregnant or nursing women
* In the presence of other ocular diseases that may affect the stability of the lens capsule (pseudoexfoliation syndrome, glaucoma, traumatic cataract, Marfan syndrome, etc.)
* Pupil abnormality (non-reactive pupil, tonic pupils, abnormally shaped pupils, etc.)
* History of any clinically significant retinal pathology or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy optic nerv atrophy, amblyopia, strabismus, microphthalmos, aniridia, epiretinal membrane etc.) in the study eyes that could alter or limit final postoperative visual prognosis.
* Patients with history of ocular trauma or prior ocular surgery including refractive procedures
* postoperative visual acuity of worse than 0.2 logMAR in any eye
* Patients using systemic or ocular medication that affect visual acuity.
* Patients participating in other clinical trials during the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bilateral cataract
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-05-31 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
monocular and binocular visual acuity | 3 months postoperatively
  uncorrected distance visual acuity (UCVA), intermediate visual acuity, near visual acuity will be measured at 5m, 80cm and 40cm respectively. All visual acuity measurements will be conducted under photopic conditions (85 cd/m2) and at 100% contrast
economic efficiency | 3 months postoperatively
  economic efficiency was defined as the ratio of objective spectacle independence (UCVA better than 0.10 logMAR) and IOL price, then compare the economic efficiency among different groups.

SECONDARY OUTCOMES:
Binocular Contrast sensitivity | 3 months postoperatively
  Contrast sensitivity measures will be conducted binocularly, under photopic, mesopic (5 cd/m2), photopic with glare and mesopic with glare conditions, with the OPTEC 6500 contrast sensitivity test (Stereo Optical, USA). Contrast sensitivity will be evaluated at five spatial frequencies (1.5, 3, 6, 12, and 18 cycles per degree [cpd]). Patients will be allowed 5 minutes to adapt to each illumination level before testing.
Binocular Defocus Curve | 3 months postoperatively
  Binocular defocus curves will be obtained in all patients, positioned at 5m under photopic (>85 cd/m 2 ) condition to measure the visual acuity with each defocus lens, representing the consecutive visual function of each eye. Negative lenses were added in 0.50 D steps and the visual acuity will be recorded for each type of defocus level. The procedure will be then repeated but with positive lenses. The range of defocus evaluated is from -4.00D to +2.00D.
stereopsis | 3 months postoperatively
  distant stereopsis will be measured by block diagram of random-spot synoptophore, while near stereopsis will be measured by Yan's stereogram.
Fusion function | 3 months postoperatively
  The fusion function of perception and movement (convergence and divergence)will be examined with a synoptophore.
Subjective visual quality | 3 months postoperatively
  Using NEI-VFQ-25 questionnaire (Chinese version). Photic phenomena, spectacle independence, and satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Hong, PhD，MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun T, Zhao X, Liu Y, Lan Q, Tang C, Qin R, Bian L, Li W, Qi H. Neurosensory binocular vision after bilateral implantation of an extended depth of focus intraocular lens with micro-monovision: a prospective cohort study. BMC Ophthalmol. 2025 May 19;25(1):294. doi: 10.1186/s12886-025-04125-5. PMID 40389895
- [Derived] Sun T, Liu Y, Gao Y, Tang C, Lan Q, Yang T, Zhao X, Qi H. Comparison of visual outcomes of a diffractive trifocal intraocular lens and a refractive bifocal intraocular lens in eyes with axial myopia: a prospective cohort study. BMC Ophthalmol. 2022 Oct 20;22(1):407. doi: 10.1186/s12886-022-02626-1. PMID 36266642
- [Derived] Lan Q, Liu Y, Xu F, Li M, Li Y, Yang T, Sun T, Yao G, Ma B, Tao L, Xiao X, Feng XL, Zeng S, Qi H. Cost-Effectiveness of Presbyopia Correction Among Seven Strategies of Bilateral Cataract Surgery Based on a Prospective Single-Blind Two-Center Trial in China. Ophthalmol Ther. 2022 Dec;11(6):2067-2082. doi: 10.1007/s40123-022-00562-3. Epub 2022 Sep 7. PMID 36071311